CLINICAL TRIAL: NCT01539876
Title: Assessing Serial Tumour Necrosis Factor Release in Locally Advanced Breast Cancer Patients Receiving Neo-adjuvant Taxane Chemotherapy
Brief Title: Tumour Necrosis Factor Release in Locally Advanced Breast Cancer Patients Receiving Neoadjuvant Docetaxel
Acronym: TNFactor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Disease Site Team changed research focus unlikely to have sufficient support to complete study
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Muriel Brackstone, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TNFactor
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
Keywords: locally advanced breast cancer patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fine Needle aspiration will be done X5: (Other): Fine Needle aspiration will be done X5: 1 hr pre-treatment, 1hr post treatment,24 hrs post treatment, 48 hrs post treatment, and following last chemotherapy cycle
  Interventions: Procedure: Fine needle aspiration assessing tumour TNFa levels

INTERVENTIONS:
Procedure: Fine needle aspiration assessing tumour TNFa levels — Fine Needle aspiration will be done X5: 1 hr pre-treatment, 1hr post treatment,24 hrs post treatment, 48 hrs post treatment, and following last chemotherapy cycle

SUMMARY:
The purpose of this study is to assess the fine needle aspiration methodology in collecting sufficient tumour cells to measure tissue TNFa levels serially in human breast cancer sample receiving Taxane treatment

DETAILED DESCRIPTION:
This pilot study will begin to test the clinical relevance of the TNFa pathway in docetaxel response in breast cancer patients receiving Taxane chemotherapy.

- Assess whether docetaxel can induce TNFa expression in breast cancer patients being treated with docetaxel

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven LABC, Locally advanced breast cancer. (operable or non-operable)
* Any T3/T4 or N2, N3 Clinical TNM stage breast cancer without metastases
* ECOG Performance Status of 0, 1 or 2.
* Patients should be able to comprehend the Letter of Information and be capable of giving informed consent.
* Female age 18 years old
* History and physical
* Negative serum pregnancy test for women of child bearing age

Exclusion Criteria:

* Inflammatory cancer (as defined by clinical evidence of dermal-lymphatic tumour involvement.)
* Ineligible for chemotherapy
* Patients with metastatic disease.
* Patients who have received prior chemotherapy or radiotherapy for this or any other malignancy.
* Previous breast cancer diagnosis
* Pregnant or lactating females are ineligible.
* Female patients of reproductive potential who decline to employ an adequate contraceptive method are ineligible.
* Participation in any concomitant trials.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
measure tissue TNFa levels | 18 months
  The TNFa levels will be evaluated using ELISA method

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Brackstone, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada